CLINICAL TRIAL: NCT03664193
Title: MRI-guided Stereotactic Body Radiotherapy (SBRT) With Simultaneous Integrated Boost for Prostate Cancer
Acronym: SIBRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802019010
Record Dates: First submitted 2018-08-30; First posted 2018-09-10 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Male patients with a histologically confirmed diagnosis of non-metastatic prostate adenocarcinoma, meeting the inclusion and exclusion criteria below, and electing to undergo definitive radiation treatment with SBRT, will be eligible for participation in this study. Patients will receive 35 Gy in five fractions, also, patients will receive a simultaneous integrated boost from 0.5-2 Gy per fx for a total dose of 37.5, 40, 42.5, or 45 Gy. Patients will also have an option to have a rectal balloon or a rectal spacer prior to receiving radiation therapy. Gastrointestinal/genitourinary toxicities will be assessed at every visit, including quality of life questionnaires and EPIC scores will be assessed at the one month follow up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): Patients will receive 35 Gy in 5 fractions. Also, patients will receive 0.5-2 Gy per fx for a total dose of 37.5, 40, 42.5, or 45 Gy. Patients will also have an option to have a rectal balloon or a rectal spacer prior to receiving radiation therapy.
  Interventions: Radiation: SIBRT

INTERVENTIONS:
Radiation: SIBRT — Patients will receive 35 Gy in 5 fractions. Also, patients will receive 0.5-2 Gy per fx for a total dose of 37.5, 40, 42.5, or 45 Gy. Patients will also have an option to have a rectal balloon or a rectal spacer prior to receiving radiation therapy.

SUMMARY:
Radiation is delivered to the prostate and seminal vesicles in 5 treatment sessions (fractions). Doses ranging from 35-45 Gy in 5 fractions have demonstrated good outcomes with acceptable toxicity.

DETAILED DESCRIPTION:
Prostate SBRT is a standard of care treatment for prostate cancer that has not spread to distant metastatic sites. Radiation is delivered to the prostate and seminal vesicles in 5 treatment sessions (fractions). Doses ranging from 35-45 Gy in 5 fractions have demonstrated good outcomes with acceptable toxicity. In this initial study, MRI guided treatment planning and delivery will be used to deliver 7 Gy to the entire prostate and seminal vesicles, with a selective boost of additional 0.5, 1.0, 1.5, or 2 Gy per fraction for a total dose of 37.5, 40, 42.5 or 45 Gy to biopsy-proven lesions, defined using MRI.

Hypothesis: MRI-guided treatment planning and delivery can selectively target high-risk prostate nodules and deliver a higher radiation dose, to achieve maximal local control without increasing treatment toxicity

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven diagnosis of prostate adenocarcinoma
2. NCCN defined low-, intermediate- and high-risk prostate cancer
3. Age ≥ 18
4. Patient must have prostate MRI with a PIRADS 3-5 lesion or PSMA positron emission tomography (PET) with an avid intraprostatic lesion

Exclusion Criteria:

1. History of prior pelvic radiation (external beam or brachytherapy)
2. Inability to undergo MRI
3. Patients with metastatic disease (other than pelvic lymph nodes) are ineligible for this study
4. American Urological Association (AUA) score >17 - AUA score >17

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with a histologically confirmed diagnosis of non-metastatic prostate adenocarcinoma, meeting the inclusion and exclusion criteria below, and electing to undergo definitive radiation treatment with SBRT, will be eligible for participation in this study.
Enrollment: 30 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Kang, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Patients will receive 35 Gy in 5 fractions. In addition, patients will also receive 0.5-2 Gy per fx for a total dose 37.5, 40, 42.5 or 45 Gy. Patients will also have an option to have a rectal balloon or a rectal spacer prior to receiving radiation therapy.
  SIBRT: Patients will receive 35 Gy in 5 fractions. In addition, patients will also receive 0.5-2 Gy per fx for a total dose 37.5, 40, 42.5 or 45 Gy. Patients will also have an option to have a rectal balloon or a rectal spacer prior to receiving radiation therapy.
Period: Overall Study
Arm/Group | Single Arm
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: Years] | 73 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 8
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Delivering Stereotactic Body Radiotherapy(SBRT) With Simultaneous Integrated Boost(SIB).
Description: Feasibility of delivering stereotactic body radiotherapy(SBRT) with simultaneous integrated boost(SIB). The investigators will track the number of treatment plans(number of participants) for each dose level (37.5, 40, 42.5, or 45 Gy) that can be delivered while meeting radiation planning objectives.
Time Frame: 2 months
Population: Patients who received stereotactic body radiotherapy(SBRT) with simultaneous integrated boost(SIB).
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Participants
  Radiation dose - 37.5Gy | 9
  Radiation Dose - 40.0Gy | 14
  Radiation Dose - 42.5Gy | 2
  Radiation Dose - 45Gy | 5
Statistical Analysis 1: Comparison: Single Arm; Test type: Other — Simple descriptive feasibility proportion and exact 95% confidence interval for radiation dose of 37.5 Gy; Proportion (percent) = 30.0, 95% CI 2-sided [14.7 to 49.3]
Statistical Analysis 2: Comparison: Single Arm; Test type: Other — Simple descriptive feasibility proportion and exact 95% confidence interval for radiation dose of 40.0 Gy; Proportion (percent) = 46.7, 95% CI 2-sided [28.3 to 65.7]
Statistical Analysis 3: Comparison: Single Arm; Test type: Other — Simple descriptive feasibility proportion and exact 95% confidence interval for radiation dose of 42.5 Gy; Proportion (percent) = 6.7, 95% CI 2-sided [0.8 to 22.1]
Statistical Analysis 4: Comparison: Single Arm; Test type: Other — Simple descriptive feasibility proportion and exact 95% confidence interval for radiation dose of 45.0 Gy; Proportion (percent) = 16.7, 95% CI 2-sided [5.6 to 34.7]

2. Primary Outcome: Number of Participants Who Received Stereotactic Body Radiotherapy(SBRT) With Simultaneous Integrated Boost (SIB) Without Greater Than Grade 3 GU/GI Toxicities.
Time Frame: 1month
Population: Patients who receive radiation dose levels of 37.5, 40, 42.5 or 45 Gy.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Participants | 30
Statistical Analysis 1: Comparison: Single Arm; Test type: Other — Simple proportion and exact 95% confidence interval; Proportion (percent) = 100, 95% CI 2-sided [88.4 to 100.0]

3. Secondary Outcome: Expanded Prostate Cancer Index Composite (EPIC) Quality of Life Questionnaires Will be Assessed in Patients.
Description: Health-related quality of life (HRQOL) measured using the Expanded Prostate Cancer Index Composite (EPIC) short-form questionnaire. The Expanded Prostate Cancer Index Composite (EPIC) is a comprehensive instrument designed to evaluate patient function and bother after prostate cancer treatment. Scores range from 0 to 100, lower scores indicate worse outcomes and higher EPIC scores represent better outcomes.
Time Frame: baseline, 3-6 months post treatment start
Population: Each time the HRQOL was administered, anywhere from 6 to 26 participants elected not to complete all the sections of the HRQOL. As such, the number of participants analyzed differs for each time point of HRQOL assessment.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline Urinary function | 87.9 [45.3 to 100]
  Baseline Bowel Function | 93.1 [50 to 100]
  Baseline Sexual function: number analyzed (Participants) | 17
  Baseline Sexual function | 58.5 [16.8 to 100]
  Baseline Hormonal Function: number analyzed (Participants) | 4
  Baseline Hormonal Function | 90 [80 to 100]
  3-6 months post - Urinary function: number analyzed (Participants) | 19
  3-6 months post - Urinary function | 93.1 [52.8 to 100]
  3-6 months post - Bowel Function: number analyzed (Participants) | 19
  3-6 months post - Bowel Function | 94.2 [54.2 to 100]
  3-6 months post - Sexual Function: number analyzed (Participants) | 17
  3-6 months post - Sexual Function | 53.3 [12.5 to 100]
  3-6 months post - Hormonal Function: number analyzed (Participants) | 7
  3-6 months post - Hormonal Function | 82.8 [80 to 100]

4. Secondary Outcome: American Urological Association (AUA) Questionnaire Will be Assessed.
Description: Health-related quality of life (HRQOL) measured using the AUA assessment will occur at baseline, and at first follow up. The American Urological Association (AUA) has developed the following questionnaire to help men determine how bothersome their urinary symptoms are and to check how effective their treatment is. 0-7 is mild, 8-19 is moderate and 20-35 is severe.
Time Frame: baseline, 3-6 months post treatment start
Population: Each time the AUA assessment was administered, anywhere from 2 to 3 participants elected not to complete all sections of the AUA assessment. As such, the number of participants analyzed differs for each time point of AUA assessment.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Single Arm
Number analyzed (Participants) | 28
score on a scale
  Baseline | 6 [1 to 14]
  3-6 month post RT: number analyzed (Participants) | 27
  3-6 month post RT | 6 [1 to 13]

ADVERSE EVENTS:
Time Frame: The adverse events were collected over a time period of 6 months.
Description: The adverse events were collected based on the CTCAEv4.03.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=30)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This event is unrelated to the study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=30)
Urinary Frequency (Renal and urinary disorders) | 23 (23)
Urinary retention (Renal and urinary disorders) | 2 (2)
Fatigue (General disorders) | 4 (4)
Urethritis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03664193/Prot_SAP_000.pdf